CLINICAL TRIAL: NCT05245981
Title: Pilot Study: Clinical Application of Mg Based Biodegradable Material for Fracture Fixation in the Adult Skeleton -First in Man Study
Brief Title: Clinical Application of Mg Based Biodegradable Material for Fracture Fixation in the Adult Skeleton
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Laura Bassi Fond; AUVA (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRI.MAG 2
Record Dates: First submitted 2022-02-02; First posted 2022-02-18 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Fracture of Medial Malleolus
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BRI.MAG 2 (Experimental): Patients presenting with dislocated isolated or combined fracture of the medialis malleolus are eligible to receive the investigational device.
  Interventions: Device: BRI.MAG 2

INTERVENTIONS:
Device: BRI.MAG 2 — Patients presenting with dislocated isolated or combined fracture of the medialis malleolus, will be screened for eligibility. Every effort will be made to ensure eligibility of the patients prior to enrollment. 20 patients will be recruited for the study.

SUMMARY:
This study is a prospective, non-randomized trial for the treatment of fractures of the medial malleolus using lean, bioabsorbable, rare-earth element (REE) free, magnesium (Mg)-based biodegradable screws in the adult skeleton.

A total of 20 patients with isolated, bimalleolar, or trimalleolar ankle fractures were recruited between July 2018 and October 2019. Fracture reduction was achieved through bioabsorbable Mg-based screws composed of pure Mg alloyed with zinc (Zn) and calcium (Ca) (0.45 wt% Zn and 0.45 wt% Ca; ZX00). Visual analogue scale (VAS) and the presence of complications (adverse events) during follow-up (12 weeks) were used to evaluate the clinical outcomes. The functional outcomes were analyzed through the range of motion (ROM) of the ankle joint and the American Orthopaedic Foot and Ankle Society (AOFAS) score. Fracture reduction and gas formation were assessed using several plane radiographs.

DETAILED DESCRIPTION:
The pilot study was designed as a prospective, nonrandomized trial for the treatment of displaced fractures of the medial malleolus with a lean, REE-free, Mg-based biodegradable implant in the adult skeleton. The trial was conducted according to the Good Clinical Practice (ISO 14155:2011) standard and the Declaration of Helsinki.The study was performed at the Department of Orthopaedics and Trauma at the Medical University of Graz and approved by the ethics committee (28 - 071 ex 15/16). A total of 20 subjects were recruited and operated on by three experienced surgeons in the centre between July 2018 and October 2019. Inclusion focused on adults aged between 18 and 65 years presenting with a displaced isolated medial malleolus fracture, a bimalleolar ankle fracture, or a trimalleolar ankle fracture. Fracture displacement was defined as diastasis of the fracture in any direction of 2 mm or more. Exclusion criteria were pathological fractures, underlying diseases (particularly bone diseases, kidney diseases, diabetes mellitus), polytraumatized patients, and pregnant or breastfeeding women.Written informed consent was obtained from each patient before the surgery. All radiological data were stored in a picture archiving and communication system (PACS). Fractures were classified according to the Herscovici system.25

Description of the bioresorbable device used: Ultra-high pure Mg (99.999%) was alloyed with Zn and Ca (0.45 wt% Zn and 0.45 wt% Ca) at 750°C under a protective gas atmosphere. Prepared screws had a length of 40 mm and a diameter of 3.5 mm. Implants were threaded at the distal part for use as traction screws.

Surgery: All patients were operated in a supine position. In case of a bimalleolar or trimalleolar fracture, the fibular and the dorsal tibial fragments were treated before the medial malleolus. Subsequently, two parallel Kirschner wires perpendicular to the medial malleolar fracture line were positioned with fluoroscopic control. A cannulated drill bit with 2.7 mm width was used for preparing the hole. Subsequently, one wire was removed and the ZX00 compression screw was inserted into the hole. Final fixation of the fracture was achieved with the second bioabsorbable Mg screw after removal of the second wire. The insertion torque of the screws was limited at a force of 1.5 newton metre with a torque handle. In all patients, no additional implants other than the Mg screws were used for the fixation of the medial malleolus. Patients with bimalleolar fractures and trimalleolar fractures were fixed with titanium plates and screws. Moreover, patients were immobilized with an under-knee plaster cast four to six weeks postoperatively and encouraged to attempt full weight-bearing as tolerated. Ankle movement exercises were started immediately after removal of the plaster.

Assessments and measurements: For each subject, the study consisted of assessments conducted preoperatively, immediately after operation and postoperative followup visits. During follow-up, complications including vital signs, erythema, swelling, pain, secretions, wound healing disorders, wound infections, or implant infections were recorded. Pain was assessed using visual analogue scale (VAS). Blood analysis and detection of Ca and Mg were recorded. Functional outcomes were evaluated through range of motion (ROM) in dorsal and plantar flexion. Additionally, the American Orthopaedic Foot and Ankle Society (AOFAS) score was performed after three months. Anteroposterior and lateral ankle radiographs (X-rays) were used to evaluate the fracture union and loss of reduction during follow-up. Postoperative radiograph evaluation was performed by two independent radiologists.

The study was registered retrospectively on Clinicaltrials.gov.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a dislocated fracture of the medial malleolus. Dislocation is defined as diastasis of the fracture in any direction of 2 mm or more.
* Otherwise healthy patients (women and men) in the age-group 18 to 65 years
* Subject has been informed of the nature of the study, agrees to participate and signs the approved consent forms. Included in this procedure is the standard information about the operation procedure.
* Subject is able and willing to comply with all assessments in the study
* Female subject with child-bearing potential perform a pregnancy test

Exclusion Criteria:

* pathological fractures (f.e. bone cyst)
* underlying diseases (particularly bone diseases, kidney diseases, diabetes mellitus)
* poly-traumatized patient
* multiple fractures at the same extremity
* pregnant or breastfeeding women
* inability or unwillingness to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Safety: Absence of (Serious) Adverse Events (SAE) throughout the study | 3 years after surgery
  (Serious) Adverse Events defined as:
  * Secondary (post-op) diastasis of the distal tibiofibular joint assessed by two plane x-rays
  * Secondary diastasis of the malleolus medialis assessed by two plane x-rays.
  * Infection of the osteosynthesis assessed clinically and/or radiologically with the presence of at least three of the following signs: clinically: pain, swelling, warmth and redness in the infected area, chills and fever x-rays: regional osteopenia, periosteal reaction/thickening, Codman's triangle, focal bony lysis, loss of bony trabecular architecture, new bone apposition
Primary Efficacy- Change of stability of the distal tibiofibular joint | after surgery, at 2 weeks and at 6 weeks
  Stability of the distal tibiofibular joint reduced with two BRI.MAG screws assessed by two plane x-rays after surgery, at 2 weeks and at 6 weeks s and at 6 weeks
Primary Efficacy- Change of stability of the fracture of the medial malleolus | after surgery, at 2 weeks and at 6 weeks
  Stability of the fracture of the medial malleolus reduced by two BRI.MAG screws assessed by two plane x-rays after surgery, at 2 weeks and at 6 weeks

SECONDARY OUTCOMES:
Procedural success - operation procedure | 6 weeks
  no change of the operation procedure from conventional to biodegradable
Procedural success- complications | 6 weeks
  Occurrence of interventional complications (break of material)

CONTACTS AND LOCATIONS:
Overall Officials: Franz Josef Seibert, Prof.Dr., Principal Investigator — Medical University of Graz, Departement of orthopaedics and traumatology
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided